CLINICAL TRIAL: NCT02912949
Title: A Phase I/II Study of MCLA-128, a Full Length IgG1 Bispecific Antibody Targeting HER2 and HER3, in Patients With Solid Tumors (eNRGy)
Brief Title: A Study of Zenocutuzumab (MCLA-128) in Patients With Solid Tumors Harboring an NRG1 Fusion (eNRGy)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Partner Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCLA-128-CL01; 2014-003277-42 (EudraCT Number)
Record Dates: First submitted 2016-08-16; First posted 2016-09-23 (Estimated); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Solid Tumours Harboring NRG1 Fusion; NSCLC Harboring NRG1 Fusion; Pancreatic Cancer Harboring NRG1 Fusion; NRG1 Fusion
Keywords: Bispecific Antibody IgG1, HER2, HER3; MCLA-128; Antibodies, Bispecific; Immunologic Factors; NRG1 fusion; Solid tumor; Pancreatic cancer; PDAC; Non-small cell lung cancer; NSCLC; zenocutuzumab
MeSH Terms: conditions — Lethal Congenital Contracture Syndrome 2; Pancreatic Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — zenocutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Part 2 Pancreatic adenocarcinoma harboring NRG1 fusion (Experimental): Participants will receive intravenous infusion of 750 mg of zenocutuzumab (MCLA-128) (the recommended Phase 2 dose (RP2D)) every 2 weeks.
  Interventions: Drug: zenocutuzumab (MCLA-128)
- Part 2 NSCLC cancer harboring NRG1 fusion (Experimental): Participants will receive intravenous infusion of 750 mg of zenocutuzumab (MCLA-128) (the recommended Phase 2 dose (RP2D)) every 2 weeks.
  Interventions: Drug: zenocutuzumab (MCLA-128)
- Part 2 Solid tumour (basket) harboring NRG1 fusion (Experimental): Participants will receive intravenous infusion of 750 mg of zenocutuzumab (MCLA-128) (the recommended Phase 2 dose (RP2D)) every 2 weeks.
  Interventions: Drug: zenocutuzumab (MCLA-128)

INTERVENTIONS:
Drug: zenocutuzumab (MCLA-128) — full length IgG1 bispecific antibody targeting HER2 and HER3
  Other Names: bispecific; MCLA-128

SUMMARY:
This is a Phase I/II, open-label, multi-center, multi-national, dose escalation, single agent study to assess the safety, tolerability, PK, PD, immunogenicity and anti-tumor activity of zenocutuzumab (MCLA-128) in patients with solid tumors harboring an NRG1 fusion (eNRGy)

DETAILED DESCRIPTION:
Study Design :

This open label (all participants know the identity of the study drug), multicenter (more than one study site), first-in-human study consisting of 2 parts. Part 1 is a dose escalation and Part 2 is a dose expansion cohort. Part 1 has been completed.

Part 2 new patient populations examine:

* Group F: Patients with NSCLC with documented NRG1 fusion
* Group G: Patients with pancreatic adenocarcinoma with documented NRG1 fusion

For these new patient populations, Part 2 will further characterize the safety and tolerability of the selected dose level of zenocutuzumab (MCLA-128), as well as assessment of CBR, defined as the proportion of patients with a CR, PR or durable SD (SD for at least 24 weeks in duration). For the new patient populations, overall response rate (ORR) and duration of response (DOR) will be described.

The study consists of 3 periods: Screening period (up to 28 days prior to the first dose of study drug); Treatment period (treatment cycles of 28 days); and Follow Up period (through 30 days after the last dose and quarterly checks for survival data for up to 2 years). Participants safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* At least one measurable lesion according to RECIST v1.1 OR evaluable disease for a limited number of patients (up to 15) in Group H;
* Performance status of ECOG 0 - 2;
* Estimated life expectancy of at least 12 weeks;
* Toxicities incurred as a result of previous anti-cancer therapy resolved to ≤Grade 1;
* Treatment with anti-cancer medication or investigational drugs within the following intervals before the first dose of MCLA-128:

  1. more than 14 days or more than 5 half-lives prior to study entry, whichever is shorter.
  2. more than 14 days for radiotherapy.
* Recovery from major surgery or other complication to ≤ Grade 2 or baseline ;
* Absolute neutrophil count ≥1.5 x 109/L without colony stimulating factor support for at least 7 days prior to screening;
* Platelets ≥75 x 109/L without transfusion support for at least 7 days prior to screening;
* Hemoglobin ≥8 g/dL or ≥5 mmol/L;
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤3 x upper limit of normal (ULN) and total bilirubin ≤1.5 x ULN; in cases of metastatic liver involvement, ALT/AST ≤5 x ULN and total bilirubin ≤2 x ULN will be allowed; in cases of antecedents of Gilbert's syndrome when total bilirubin ≤3.0 x ULN or direct bilirubin ≤1.5 x ULN will be allowed;
* Estimated glomerular filtration rate (GFR) of more than 30 mL/min
* Able to provide a tumor biopsy sample (fresh strongly preferred or else archival);
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 6 month after completion of study therapy;
* Patients must have received prior standard therapy appropriate for their tumor type and stage of disease, or in the opinion of the Investigator, would be unlikely to tolerate or derive clinically meaningful benefit from appropriate standard of care therapy or no satisfactory alternative treatment options are available;
* Locally-advanced unresectable or metastatic solid tumor malignancy with documented NRG1 gene fusion, identified through molecular assays such as next generation sequencing-based assays [DNA or RNA], as routinely performed at CLIA or other similarly-certified laboratories.

Exclusion Criteria:

* Pregnant or lactating;
* Presence of an active uncontrolled infection or an unexplained fever;
* Known hypersensitivity to any of the components of MCLA-128;
* Known HIV, active Hepatitis B without receiving antiviral treatment, or Hepatitis C; patients treated for Hepatitis C and have undetectable viral loads are eligible
* Known symptomatic or unstable brain metastases;
* Patients with leptomeningeal metastases;
* Presence of LVEF below 50% on the screening echocardiogram; or history or presence of any significant cardiovascular disease, including unstable angina or myocardial infarction within 12 months prior to screening, congestive heart failure (NYHA Class III or IV), or ventricular arrhythmia requiring medication;
* Previous or concurrent malignancy (excluding non-basal cell carcinoma of skin or carcinoma in situ of the uterine cervix) unless the tumor was treated with curative intent more than 2 years prior to study entry;
* Presence of any other medical or psychological condition deemed by the Investigator to be likely to interfere with a patient ability to sign informed consent, cooperate or participate in the study, or interfere with the interpretation of the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective overall response rate (ORR) as per local investigator's assessment | 36 months
  Evaluation of clinical benefit assessed by RECIST v1.1 determining objective overall response rate (ORR)
Duration of response per RECIST v1.1 as per local Investigator's assessment. | 36 Months
  To assess durability of anti-tumor activity of MCLA-128 in patients with NRG1 fusions as assessed locally

SECONDARY OUTCOMES:
Overall response rate as per Blinded Independent Central Review (BICR) | 36 months
  Assess the anti-tumor response of zenocutuzumab (MCLA-128) by RECIST v1.1 as assessed centrally
Clinical Benefit Rate (CBR) of zenocutuzumab (MCLA-128) assessed locally and BICR | 36 months
  CBR assessed as the proportion of patients in whom a complete response (CR) or partial response (PR) or stable disease (SD) is observed (where SD duration is a minimum of 24 weeks) by RECIST v1.1 .
Duration of Response as per BICR | 36 months
  To assess durability of anti-tumor activity of MCLA-128 in patients with NRG1 fusions as assessed centrally
Time to response per RECIST v1.1. as per local investigator assessment | 36 months
  To assess time to onset of response in patients with NRG1 fusions as assessed locally
Time to response per RECIST v1.1. as per BICR | 36 months
  To assess time to onset of response in patients with NRG1 fusions as assessed centrally
Characterize the safety and tolerability of zenocutuzumab (MCLA-128) | 6-12 months
  Number of participants with Adverse Events (AE) and Serious Adverse Events (SAE)
Maximum plasma concentration [Cmax] | 36 months
  Assess the Cmax of zenocutuzumab (MCLA-128)
Volume of distribution [V] | 36 months
  Assess the volume of distribution of zenocutuzumab (MCLA-128)
Volume of distribution at steady state [Vss] | 36 months
  Assess the volume of distribution of zenocutuzumab (MCLA-128) at steady state
Area under the concentration versus time curve from time zero to time t [AUC0-t] | 36 months
  Assess the Area under the concentration versus time curve from time zero to time t [AUC0-t] of zenocutuzumab (MCLA-128)
half-life [t1/2] | 36 months
  Assess the half-life of zenocutuzumab (MCLA-128)
area under the concentration versus time curve [AUC0-∞] | 36 months
  Assess the area under the concentration versus time curve [AUC0-∞] of zenocutuzumab (MCLA-128)
time to reach maximum concentration [tmax] | 36 months
  Assess the time to reach maximum concentration [tmax] of zenocutuzumab (MCLA-128)
Incidence of anti-drug antibodies against zenocutuzumab (MCLA-128) | 36 months
  Assess the Incidence of anti-drug antibodies against zenocutuzumab (MCLA-128)
serum titers of anti-drug antibodies | 36 months
  Assess serum titers of anti-drug antibodies
Evaluation of progression free survival (PFS) | 36 months
Evaluation of overall survival (OS) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alison Schram, MD, Principal Investigator — Memorial Sloan Kettering Medical Center
Locations (64):
- United States (26):
  - Mayo Clinic, Phoenix, Arizona
  - The Oncology Institute of Hope and Innovation, Cerritos, California
  - University of California Irvine, Irvine, California
  - Stanford University, Palo Alto, California
  - Sharp Memorial Hospital, San Diego, California
  - Georgetown University, Washington D.C., District of Columbia
  - Memorial Cancer Institute, Hollywood, Florida
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Emory Winship Cancer Institute, Atlanta, Georgia
  - Northwest Oncology & Hematology, Rolling Meadows, Illinois
  - Dana Farber Cancer Center, Boston, Massachusetts
  - Karmanos Cancer Center, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Billings Clinic Cancer Center, Billings, Montana
  - St. James Healthcare, Butte, Montana
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Averra Medical Group, Sioux Falls, South Dakota
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Hematology-Oncology Specialist of Fredericksburg, Fredericksburg, Virginia
  - Virginia Mason Hospital & Seattle Medical Center, Seattle, Washington
  - Hematology Oncology Associates, Spokane, Washington
  - Northwest Medical Specialties, Tacoma, Washington
- Salzburger Universitatsklinikum, Salzburg, Austria
- UZ Leuven, Leuven, Belgium
- Princess MargaretCancer Centre, Toronto, Ontario, Canada
- Rigshospitalet, Copenhagen, Denmark
- France (5):
  - Centre Leon Berard, Lyon
  - Hospital Louis Pradel, FR, Lyon
  - Institut Gustave Roussy, Paris
  - Hopital Cochin, Paris
  - Hopital Curie, Paris
- Germany (3):
  - Asklepios Klinik Altona, Hamburg
  - Asklepios Kliniken Hamburg GmbH, Hamburg
  - Deutsches Krebsforschungszentrum, Heidelberg
- Israel (2):
  - Shaare Zedek Medical Center, Jerusalem
  - Sheba Medical Center, Tel Aviv
- Italy (3):
  - Niguarda Cancer Centre, Milan
  - Ospedale San Raffaele, Milan
  - Istituti Fisioterapici Ospitalieri, Roma
- Japan (4):
  - National Cancer Center Hospital, Chūōku
  - St. Marianna University School of Medicine Hospital, Kawasaki
  - Osaka International Cancer Institute, Osaka
  - National Cancer Center East, Tokyo
- Netherlands (3):
  - NKI, Amsterdam
  - Amsterdam Medical Center, Amsterdam
  - Radboud University Medical Center, Nijmegen
- University Hospital Oslo, Oslo, Norway
- National Cancer Centre of Singapore PTE LTD, Singapore, Singapore, Singapore
- South Korea (3):
  - Samsung Medical Center, Seoul
  - Seoul National University College of Medicine, Seoul
  - Severance Hospital- Yonsei Cancer Center, Seoul
- Spain (6):
  - Vall D'Hebron Institute of Oncology (VHIO), Barcelona
  - START Hospital Fundación Jiménez Diaz, Madrid
  - START Hospital Universitario Madrid Sanchinarro, Madrid
  - Hospital 12 de Octubre, Madrid
  - Clínica Universidad de Navarra, Pamplona
  - Instituto Valenciano Oncologia, Valencia
- Karolinska Universitetssjukhuset, Solna, Sweden
- National Taiwan University Hospital 7, Taipei, Taiwan
- Sarah Cannon Research Institute, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schram AM, Goto K, Kim DW, Macarulla T, Hollebecque A, O'Reilly EM, Ou SI, Rodon J, Rha SY, Nishino K, Duruisseaux M, Park JO, Neuzillet C, Liu SV, Weinberg BA, Cleary JM, Calvo E, Umemoto K, Nagasaka M, Springfeld C, Bekaii-Saab T, O'Kane GM, Opdam F, Reiss KA, Joe AK, Wasserman E, Stalbovskaya V, Ford J, Adeyemi S, Jain L, Jauhari S, Drilon A; eNRGy Investigators. Efficacy of Zenocutuzumab in NRG1 Fusion-Positive Cancer. N Engl J Med. 2025 Feb 6;392(6):566-576. doi: 10.1056/NEJMoa2405008. PMID 39908431
- [Derived] Kim DW, Schram AM, Hollebecque A, Nishino K, Macarulla T, Rha SY, Duruisseaux M, Liu SV, Al Hallak MN, Umemoto K, Wesseler C, Cleary JM, Springfeld C, Neuzillet C, Joe A, Jauhari S, Ford J, Goto K. The phase I/II eNRGy trial: Zenocutuzumab in patients with cancers harboring NRG1 gene fusions. Future Oncol. 2024;20(16):1057-1067. doi: 10.2217/fon-2023-0824. Epub 2024 Feb 13. PMID 38348690
- See also: For more information about MCLA-128 and the MCLA-128-CL01 study — http://www.nrg1.com